CLINICAL TRIAL: NCT06974045
Title: Evaluation of a Single-stage Laparoscopic Cholecystectomy and Laparoscopic Common Bile Duct Exploration Service Pre-, Intra- and Post-COVID-19 Pandemic: a Retrospective Cohort Study
Brief Title: Impact of COVID-19 Pandemic on Single-stage Laparoscopic Cholecystectomy and Laparoscopic Common Bile Duct Exploration Service
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: HH2025
Record Dates: First submitted 2025-05-13; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Gallstone
MeSH Terms: conditions — Gallstones

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

GROUPS / COHORTS (3):
- Pre-pandemic: April 2016 to March 2020 (48 months)
  Interventions: Other: Single-stage LC + LCBDE
- Intra-pandemic: March 2020 to December 2021 (22 months)
  Interventions: Other: Single-stage LC + LCBDE
- Post-pandemic/recovery period: January 2022 to February 2024 (26 months)
  Interventions: Other: Single-stage LC + LCBDE

INTERVENTIONS:
Other: Single-stage LC + LCBDE — Choledochotomy and transductal common bile duct exploration or transcystic choledochoscopy and common bile duct exploration

SUMMARY:
Choledocholithiasis is reported to be present in 15-20% of patients with symptomatic gallstones. The single-stage management consists of performing either laparoscopic common bile duct exploration (LCBDE) or intraoperative endoscopic retrograde cholangiopancreatography (ERCP) at the same time as laparoscopic cholecystectomy (LC).

Since the Coronavirus (COVID-19) pandemic, surgical practice has significantly been impacted. The pandemic has had ramifications on patient and staff safety, surgical techniques, minimally invasive procedures, theatre workflow, education and training.

We analysed a series of LCBDE procedures in our institution pre-, intra- and post-COVID-19 pandemic to assess the feasibility, efficacy and safety of this single-stage treatment approach following the pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Patients that underwent single-stage LC + LCBDE for the management of choledocholithiasis with concomitant gallstones.

Exclusion Criteria:

* Patients that underwent LC only or LCBDE only

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients that underwent the single-stage approach of LC + LCBDE for the management of choledocholithiasis, between April 2016 and February 2024. All patients were assessed with preoperative liver function tests (LFTs) and abdominal imaging such as ultrasound, computed tomography (CT) and/ or magnetic resonance cholangiopancreatography (MRCP).
Sampling Method: Non-Probability Sample
Enrollment: 237 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Intraoperative measures | 90 days
  Size of choledochoscope, holmium laser lithotripsy use and stone clearance rates
Postoperative complications | 90 days
  Complications such as bile leak and pancreatitis, including hospital length of stay